CLINICAL TRIAL: NCT03859817
Title: Observational Study to Evaluate the Relationship Between Ketonemia and Renal Function in the Diabetic Patient
Acronym: TAKEN-DKD
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Paolo Fiorina, MD, Clinical Professor, University of Milan
Other Study IDs: 2018/ST/043
Record Dates: First submitted 2019-02-28; First posted 2019-03-01 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Diabetic Nephropathy Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples Without DNA — Collection of blood sample for immunological study (blood sampling to be performed on fasting) Urine sample collection for immunological study (collection carried out on the day of the visit)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with albuminuria: Comparison of eGFR values and ketonemia in diabetic patients
  Interventions: Other: Comparison of eGFR values and ketonemia in diabetic patients
- patients with normo albuminuria: Comparison of eGFR values and ketonemia in diabetic patients
  Interventions: Other: Comparison of eGFR values and ketonemia in diabetic patients

INTERVENTIONS:
Other: Comparison of eGFR values and ketonemia in diabetic patients — To verify if there is a correlation between the level of ketones and an alteration of the renal function in the diabetic patient, the values of the prognostic markers indicated in the protocol and the data downloaded by the glucometers will be evaluated in addition to the blood tests of the patients

SUMMARY:
A multicentre real life study is proposed. The study has as its goal primary to compare the levels of ketonemia measured in patients with albuminuria and patients normo albuminurici to evaluate a possible correlation between ketone level and alteration of renal function in the diabetic patient, comparing the eGFR values of patients with ketonemia high and of patients with low ketonemia. In these patients, the lack of insulin causes one imbalance between ketogenesis and ketolysis, with increased production and reduced body clearance ketones. Several studies explore the effects of ketone bodies on cell function and lesions diabetic complications: ketonemia induces oxidative stress and increases the risk and the progression of complications, moreover, the increase in ketone levels may have pro-inflammatory effects. However, ketonemia levels between normal and DKA are poorly studied and their effects are still unknown. It is hypothesized that

* in diabetic patients with DKD the level of ketones may be high;
* Increased ketone levels may promote an alteration of renal function.

We want to evaluate the relationship between ketone levels and renal function, because the kidneys, as well as the heart, are among the main organs in which the ketone bodies are oxidized to produce energy and DKD has a high morbidity and mortality in diabetes. The main objectives for being able to demonstrate the hypothesis in question are:

* Evaluate the level of ketones in albuminurate patients with diabetes and in patients with renal function altered;
* Evaluate the association between ketone level and decline of renal function in the diabetic patient e therefore the impact of ketonemia on the progression of renal function loss.

DETAILED DESCRIPTION:
At the beginning and during the course of the study the glycemic and ketone index obtained by the homologous blood glucose monitoring will be evaluated. During the study, prognostic biomarkers (sP2X7R, KIM-1, sTNFR1, 11-dehydro-tromoxane B2 and 6-keto-prostaglandin-F-1a (PGF1α)), which are presumed to play an important role in inflammatory renal diseases, will also be measured in diabetic subject, in addition to the traditional marker that is the urinary albumin.

Step 1. Visit Baseline: blood sampling and collection of a urinary sample, evaluation proteinuria, GFR and blood and urinary ketones Step 2. Visit at 6 months: blood collection and collection of a urinary sample, evaluation proteinuria, GFR and blood and urinary ketones Step 3. Visit at 12 months: blood collection and collection of a urinary sample, evaluation proteinuria, GFR and blood and urinary ketones. The study involves the enrollment of T1D and T2D subjects in diabetic nephropathy. The study involves the enrollment of T1D and T2D subjects in diabetic nephropathy A timetable will be prepared for the surgeries during the which the diabetic subject will be informed about the study protocol in question and will provide eventual informed consent to entry into the study, blood sampling and urinary sample collection. However, the analysis will be above all exploratory and will allow to foresee possible studies future properly sized.

ELIGIBILITY:
Inclusion Criteria:

Presence of albuminuria (≥30 mg / 24h)

* Adult and male patients of age
* Diagnosis of type 1 or type 2 diabetes according to the ADA diagnostic criteria
* Presence of the disease for at least five years
* HbA1c≥7%
* Written informed consent of the patient and / or parents or legal guardian

Exclusion Criteria:

Chronic end-stage renal disease (CKD5)

* Current or previous treatments with immunosuppressants (with the exception of topical steroids ed inhalers)
* Participation in other clinical studies
* Significant disease other than diabetes found in the two weeks prior to the first visit
* Neurological or psychiatric diseases, hemoglobinopathies, liver diseases, cancer, cystic fibrosis, renal failure, malabsorption syndromes
* Abuse of alcohol and drugs
* HIV or hepatitis
* Pregnant or lactating women (β-HCG urinary should be evaluated before each visit)
* Presence of serious diseases or conditions of the patient considered unsuitable by the Investigator for be able to include it in the study
* Poor understanding by the patient of spoken and written Italian

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited based on anamnestic and clinical data and blood and urine parameters specific for type 1 diabetes mellitus and type 2 diabetes mellitus in diabetic nephropathy.
Sampling Method: Probability Sample
Enrollment: 68 (Estimated)
Dates: Start 2019-04-16 (Actual); Primary Completion 2021-12-18 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Variations in albuminuria and albumin / creatinine ratio in urine (UACR) | 12 months
  immunoturbidimetric method
Variations of the eGFR (CKD-EPI formula) | 12 months
  CKD-EPI formula
Variations in ketone levels | 12 months
  monitoring ketones in capillary and urinary samples

SECONDARY OUTCOMES:
Variations of tubular function markers (sP2X7R, KIM-1, sTNFR1) | 12 months
  enzyme immunoassay (ELISA)
Variations of markers of glomerular function (11-dehydro-tromoxane B2 and 6-keto-prostaglandin- F-1a (PGF1α)) | 12 months
  enzyme immunoassay (ELISA)
Changes in glycated hemoglobin (HbA1c) | 12 months
  capillary electrophoresis

CONTACTS AND LOCATIONS:
Locations (1):
- ASST FBF-Sacco P.O. Sacco/Fatebenefratelli e Oftalmico, Milan, Italy